CLINICAL TRIAL: NCT05991414
Title: The Effect of Pharmacist-Initiated Home Blood Pressure Monitoring on Blood Pressure Control in Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00128951
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Participants in Control Group will be offered opportunity to crossover to the Intervention Protocol after their initial 6-month study period.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacist care in conjunction with home blood pressure monitoring (Experimental): Patients will have BP assessed at baseline in the pharmacy by the pharmacist, and they will receive a home blood pressure monitor in addition to education and counselling provided by the pharmacist. Patients will measure their BP at home for seven days every four weeks and input their results into a data management system called REDCap that is accessible by the pharmacist. The pharmacist will follow up with the patient every 4 weeks to review their readings and at 24-weeks the patient will come into the pharmacy for a final follow-up and BP readings. The pharmacist will fax BP readings as well as suggestions for therapy modification to the patient's prescribing clinician. Patients will then have their care returned to their prescribing clinician with no pharmacist specific interventions outside of usual pharmacy care activities and have a single follow-up at month-12 with the pharmacist reviewing home BP monitor use and reporting of data to prescribing clinician.
  Interventions: Device: Home blood pressure monitor; Procedure: Enhanced community pharmacist care
- Usual pharmacist care (Active Comparator): Patients will have BP assessed at baseline, 12-, and 24-weeks in the pharmacy by the pharmacist. Patients will not receive a home blood pressure monitor. Pharmacist will provide them usual care, education and counselling on BP management. Pharmacists will fax BP readings to the patient's prescribing clinician but will not provide any suggestions for therapy modification. After 24-weeks patients will be offered a home blood pressure monitor with education on its use. They will then be offered to crossover to the intervention group for the next 6-months or have their care returned to their prescribing clinician with no pharmacist specific interventions outside of usual pharmacy care activities and have a single follow-up at month-12 with the pharmacist reviewing home BP monitor use and reporting of data to prescribing clinician.
  Interventions: Procedure: Usual pharmacist care

INTERVENTIONS:
Device: Home blood pressure monitor — Participants provided home blood pressure monitor and instructions on use from pharmacist. They will measure home BP every 4-weeks for 7 days as per Hypertension Canada 7-day home BP protocol.
  Arms: Pharmacist care in conjunction with home blood pressure monitoring
Procedure: Enhanced community pharmacist care — Pharmacist to follow up with participants every month to review home BP readings. Then the pharmacist will send home BP readings and recommendations for changes to antihypertensive medication regimen to participants prescribing clinician. Pharmacist will then advise participants to follow up with their prescribing clinician.
  Arms: Pharmacist care in conjunction with home blood pressure monitoring
Procedure: Usual pharmacist care — Participants will come into the pharmacist at baseline, 12- and 24-weeks to have their BP taken by the pharmacist. Pharmacist will provide education and counseling. Pharmacist will send BP readings to participants prescribing clinician with no recommendations for changes to antihypertensive therapy. After 6-months participants will be offered a home BP monitor and instructions on use.
  Arms: Usual pharmacist care

SUMMARY:
To evaluate the impact of home blood pressure monitoring when used in addition to pharmacist care, compared to usual care, in women with elevated blood pressure (BP). Randomized 1:1 two-arm controlled trial. Patients to be identified and screened by pharmacists. Patients with a BP >140/90mmHg or >130/80mmHg in those with diabetes will be invited to enroll in the study.

Intervention: Patients will have BP assessed at baseline by the pharmacist, and they will receive a home blood pressure monitor in addition to counselling provided by the pharmacist. Patients will measure their BP at home for seven days every four weeks and input their results into a data management system. The pharmacist will follow up with the patient every 4 weeks to review their readings and at 24-weeks the patient will come into the pharmacy for a final follow-up and BP readings. The pharmacist will fax BP readings and suggestions for therapy modification to the patient's prescribing clinician. After 24-weeks patient care is returned to the prescribing clinician with no further pharmacist interventions except for a final post-trial follow-up at week-52 to review ongoing home BP monitor use and BP management by the prescribing clinician.

Control: Patients will have BP assessed at baseline, 12-, and 24-weeks in the pharmacy by the pharmacist. Patients will not receive a home blood pressure monitor. Pharmacist will provide usual care, education and counselling on BP management. Pharmacists will fax BP readings to the patient's prescribing clinician but will not provide any suggestions for therapy modification. After 24-weeks patients will be offered a home blood pressure monitor with education on its use. They will then be offered to crossover to the intervention group for the next 24-weeks or have their care returned to their prescribing clinician with no pharmacist specific interventions except for a final post-trial follow-up at week-52 to review ongoing home BP monitor use and BP management by the prescribing clinician.

Sample Size: Calculated sample size is 368 participants to achieve 80% power, with 184 patients in the intervention and control groups.

Primary Outcome: Difference in change in Systolic Blood Pressure between the home blood pressure monitoring in addition to pharmacist care versus usual care group.

DETAILED DESCRIPTION:
Purpose:

To determine the impact of home blood pressure monitoring when used in addition to pharmacist care, compared to usual care, in women with blood pressure elevated above their target level.

Hypothesis:

Women patients utilizing home blood pressure monitors and providing blood pressure readings to their community pharmacists who then provides tailored education to the patient and therapy recommendations to the patient's prescribing clinician will result in greater improvements in blood pressure control. In comparison to usual care.

Justification:

* Women are a target population for blood pressure control. A majority of women in Canada are not achieving their target blood pressure for optimal health outcomes.
* Home blood pressure monitors have demonstrated benefit in supporting patients in reaching their blood pressure targets, although they are under utilized.
* Community pharmacist care also has demonstrated benefit in supporting patients in reaching their blood pressure targets.
* Community pharmacies are where patients can acquire a home blood pressure monitor.

Research Method and Procedures:

Randomized Controlled Trial - Study length is 24-weeks with a final follow-up at 52-weeks.

Study Setting: Community Pharmacies throughout Ontario, Canada. Pharmacies will be selected identified and selected based on their location, using definitions of urban and rural communities from Statistics Canada's Statistical Area Classifications, and their willingness to partake in the study itself and follow-up with participants. The study is aiming to recruit a 50:50 ratio of pharmacies from urban and rural communities.

Screening/Case Finding:

Pharmacists may identify potential participants for screening via the following methods:

* During their usual workflow in providing patient care.
* During a hypertension screening day at the pharmacy.
* Searching patient pharmacy profiles with the following medication classes: Antidiabetes, antiobesity, antianginals, antihypertensive, cholesterol-lowering, smoking cessation therapies, prenatal vitamins or commonly used antihypertensives used during pregnancy such as methyldopa or labetalol.
* Referral from another healthcare provider.

Recruitment:

Once screening is complete if the participant is eligible for participation they will be asked by the pharmacist to provide consent. Consent will be obtained electronically via the REDCap database management system. Once consent is obtained the participant will be enrolled in the study and randomized to one of the two groups using the REDCap randomization module.

Both Groups:

* Pharmacist will measure participants blood pressure in the pharmacy using a standardized method based on the technique described by Hypertension Canada.
* Each participating pharmacy will be provided with a BIOS BD270 Automated Office Blood Pressure Monitor.
* Data to be collected by the pharmacist and input by the participant at baseline and week-24 includes demographics, medical history, medications, social history and cardiovascular risk factors.
* Participants prescribing clinician will be informed about the participants enrolment in the study.

Intervention Group:

* AOBP readings in the pharmacy will be taken at baseline and week-24.
* Participants will be provided with a BIOS BD240 home blood pressure monitor. Participants will measure their blood pressure at home every four weeks for five four week periods - they will take two consecutive BP readings in the morning and in the evening for a period of 7-days as per the Hypertension Canada 7-day BP Protocol. Participants will upload their data into the REDCap database via digital links sent via text message or email.
* Pharmacist will review BP readings with the participant at baseline and every 4 weeks. They will also send the BP readings along with suggestions for therapy modification to the participants prescribing clinician.
* After 24-weeks care is returned to the prescribing clinician and no further pharmacist specific interventions will be provided. The primary study will be complete at this point.
* After 52-weeks the pharmacist will complete a final follow-up to assess ongoing use of home blood pressure monitor and if there had been any further interactions with the prescribing clinician. No further follow-ups in regards to the study will occur beyond this point.

Control Group:

* AOBP readings in the pharmacy will be taken at baseline, week-12 and week-24.
* Participants will not be provided with a home blood pressure monitor.
* Pharmacists will review BP readings with the participant at each follow up and they will send BP readings to the participants prescribing clinician. The pharmacist will provide no recommendations for therapy modification.
* After the week-24 follow up participants will be offered a BIOS BD240 home blood pressure monitor. They will also be offered the opportunity to crossover to the intervention group for the next 24-weeks. If the participant agrees to crossover they will receive the full intervention protocol with the exception of the final follow-up at week-52. If they decline to crossover care is returned to the prescribing clinician and no further pharmacist specific interventions will be provided. The primary study will be complete at this point. After 52-weeks the pharmacist will complete a final follow-up to assess ongoing use of home blood pressure monitor and if there had been any further interactions with the prescribing clinician. No further follow-ups in regards to the study will occur beyond this point.

Sample Size:

Calculated to be 320 participants to achieve 80% power. This assumes an estimated SD of 13.5 to detect a difference in change of AOBP Systolic Blood Pressure of 4.5mmHg. We have assumed a drop-out or loss to follow up rate of 15% which increases our sample size to 368 participants with 184 participants in each group.

Plan for Data Analysis:

Data will be collected in the RedCap Database. Data will be analyzed in conjunction with the ABSPOR Unit who is providing the support for data analysis, interpretation and data visualization.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included if they are female ≥18 years of age and meet one of the following criteria:

No established diagnosis and/or treatment for hypertension.

* Average of three AOBP readings at two pharmacy visits within a 2-week period:
* SBP ≥140 mmHg or DBP ≥90 mmHg
* SBP ≥130 mmHg or DBP ≥80 mmHg if they have diabetes

Established diagnosis or currently on treatment for hypertension.

* Average of three AOBP readings from one pharmacy visit:
* SBP ≥140mmHg or DBP ≥90mmHg
* SBP ≥130mmHg or DBP ≥80mmHg if they have diabetes

Exclusion Criteria:

* Male
* Having hypertensive urgency or emergency as determined on screening defined as (these patients will be referred to urgent care):
* Severe elevation of SBP >180mmHg and/or DBP >120mmHg
* Taking oral contraceptives
* Arm that <24cm (9.4") or an arm that is >43cm (17")
* Currently have, or are using a home blood pressure monitor
* No access to a smartphone or internet
* Unwilling or unable to participate or provide informed consent and sign the consent form
* If the patient is pregnant
* Participating or planning to participate in another research study or project

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference in change in Systolic Blood Pressure | 24-weeks
  Difference in change in Systolic Blood Pressure between the home blood pressure monitoring in addition to pharmacist care versus usual care group.

SECONDARY OUTCOMES:
Proportion at BP target | 24-weeks
  Proportion of patients at their BP target at 24-weeks, compared between intervention and control groups.
Percentage of home blood pressure readings recorded | 24-weeks
  Percentage of HBPM readings input by patients in the intervention groups each month during the 7-Day BP Monitoring protocol. This will be reported as a percentage of the expected measurements which is 28 inputs each month.
Adherence to Medications | 24-weeks
  Participants will be asked at each follow-up:
  Number of doses missed or forgotten between follow-up periods. The medication that the participant missed or forgot to take will be noted.
Changes to antihypertensive medication regimen | 24-weeks
  Number of new antihypertensive medications that are initiated and compared between groups.
  Number of antihypertensive medication changes and compared between groups. Number of antihypertensive dosage changes (increases or decreases) and compared between groups.
Lifestyle changes | 24-weeks
  Number lifestyle changes made by a patient, such as increased activity, smoking cessation, self-reported weight-loss, reduced intake of salt and processed foods.
Consultant Satisfaction | 24-weeks
  Patient's general satisfaction with pharmacist care measured by Consultant Satisfaction questionnaire and compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Tsuyuki, PharmD, Principal Investigator — University of Alberta
Locations (26):
- Canada (26):
  - Hills Clinic Pharmacy, Aylmer, Ontario
  - Eagle Ridge Pharmacy, Barrie, Ontario
  - Mcintyre IDA, Blenheim, Ontario
  - Shopper's Drug Mart #646, Collingwood, Ontario
  - Trailside Pharmacy Pharmasave, Fergus, Ontario
  - Health Care Pharmacy Pharmasave 683, Greater Sudbury, Ontario
  - HealthMax Pharmacy, Hamilton, Ontario
  - Inverary Pharmasave, Kingston, Ontario
  - Kawartha Lakes Pharmacy, Lindsay, Ontario
  - Guardian MarkhaMack Pharmacy, Markham, Ontario
  - Zak's Pharmacy, Milton, Ontario
  - Custom Health Pharmacy, Mississauga, Ontario
  - Sav-ON IDA Pharmacy, Oakville, Ontario
  - Lifecare Rx Pharmacy, Oakville, Ontario
  - Countryside Pharmacy, Omemee, Ontario
  - The Medicine Shoppe Pharmacy #143, Ottawa, Ontario
  - Brisson Pharmacy, Ottawa, Ontario
  - Pharmasave Sally's Pharmacy, Owen Sound, Ontario
  - Kashyaps Pharmacy Peterborough, Peterborough, Ontario
  - Port Weller Pharmacy, Saint Catherines, Ontario
  - Hogan at the Bluewater Medical Clinic, Sarnia, Ontario
  - Medicine Shopper #297, Scarborough Village, Ontario
  - Springwater Pharmacy, Springwater, Ontario
  - Shopper's Drug Mart #500, Toronto, Ontario
  - Shopper's Drug Mart #994, Toronto, Ontario
  - Ultima Apothecary, Windsor, Ontario

IPD SHARING:
Plan to Share IPD: No